CLINICAL TRIAL: NCT05296590
Title: Monocyte Distribution Width (MDW) in the General Population of Emergency Department Patients With and Without Bacteremia
Status: Active, not recruiting | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Beckman Coulter, Inc. (Industry)
Responsible Party: Principal Investigator, Anja Kathrin Jaehne, Clinical Research Coordinator, Henry Ford Health System
Other Study IDs: 14940
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Bacteremia; Bacteremia Sepsis; Sepsis; Septic Shock; Severe Sepsis; Emergency Departments; Continuity of Patient Care
Keywords: Blood Stream Infection; BSI; Bacteremia; Sepsis; Severe Sepsis; Septic Shock; Emergency Departments; Continuity of Patient Care
MeSH Terms: conditions — Bacteremia; Sepsis; Shock, Septic; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Positive Blood Culture/ Monocyte Distribution Width Normal: No intervention Monocyte Distribution Width considered normal (MDW less than 20 IU) in Emergency Department patients with Positive Blood Cultures.
  We will evaluate associated factors with this observation.
  Interventions: Diagnostic Test: Monocyte Distribution Width (MDW) , observation
- Positive Blood Culture/ Monocyte Distribution Width Abnormal: No intervention Monocyte Distribution Width considered abnormal (MDW equal or greater than 20 IU) in Emergency Department patients with Positive Blood Cultures.
  We will evaluate associated factors with this observation.
  Interventions: Diagnostic Test: Monocyte Distribution Width (MDW) , observation
- Negative Blood Culture/ Monocyte Distribution Width Normal: No intervention Monocyte Distribution Width considered normal (MDW less than 20 IU) in Emergency Department patients with negative Blood Cultures.
  We will evaluate associated factors with this observation.
  Interventions: Diagnostic Test: Monocyte Distribution Width (MDW) , observation
- Negative Blood Culture/ Monocyte Distribution Width Abnormal: No intervention Monocyte Distribution Width considered abnormal (MDW equal or greater than 20 IU) in Emergency Department patients with negative Blood Cultures.
  We will evaluate associated factors with this observation.
  Interventions: Diagnostic Test: Monocyte Distribution Width (MDW) , observation

INTERVENTIONS:
Diagnostic Test: Monocyte Distribution Width (MDW) , observation — Observation of MDW performance blinded to treating clinical teams

SUMMARY:
This project will evaluate the usefulness of Monocyte Distribution Width (MDW) for the diagnosis of blood culture positivity (BSI) in patients in the Emergency Department (ED) and reevaluate the usefulness of MDW in patients with BSI and sepsis. Consequently, if MDW indicate a high likelihood of bacteremia antibiotic management in patients with suspected bacterial infections will be changed and aid appropriate antibiotic administration.

DETAILED DESCRIPTION:
BIOMARKERS for Sepsis and Infection should address important clinical aspects such as

1. Rapid diagnosis of invasive infections contributing to organ dysfunction;
2. Provide information regarding antibiotic susceptibility and
3. Distinguish infection mediated organ dysfunction from non-infectious sepsis mimics.

Review of MDW values for ED patients who have positive blood cultures The gold standard for the diagnosis of bloodstream infections is positive blood cultures. Not all patients with sepsis have positive blood cultures, however patients with blood stream infections and end-organ dysfunction are septic and need to be treated with antibiotics. Two definitions of sepsis currently are used.

The sepsis-2 definitions [1,2] are based on a confirmed or suspected infectious source, a systemic response with two or more abnormal systemic inflammatory response syndrome criteria such as hyper or hypothermia, tachycardia, tachypnea and leukopenia or leukocytosis or bandemia and signs of at least one new end organ dysfunction. There is a differentiation between different degrees of disease severity between sepsis, severe sepsis and septic shock. Each of these degrees of illness severity are associated with different morbidity and mortality.

The sepsis-3 definition [3] state that sepsis is the bodies response to an infectious agent. The response is assessed using a quick SOFA score (qSOFA) assessment based on tachypnea of equal or greater than 22 breath, systolic hypotension of equal or less than 100 mmHg and changes in mentation measured by a Glasgow Coma Score (GCS) of less than 15 along with the requirement of a new onset of organ dysfunction as measured by a SOFA score of equal or greater than 2.[4] Sepsis-3 definition distinguish between sepsis and septic shock only. Septic shock is only present if a patient has 2 or more qSOFA criteria, requires the use of a vasoactive agent to maintain a mean arterial blood pressure of 70 mmHg AND if the lactate is greater than 2 mg/dL. Patients which do not have a qSOFA score of greater than 2 or a SOFA score of less than 2 are considered not septic and as having only a local infection.

Both definitions have the requirement for a proven or suspected infection. Source identification is important, however not always successful. The most common site of infection is the lung. This infection is most commonly viral or bacterial. The second most common site of infection is the genitourinary tract followed by blood stream infections. The diagnosis of blood stream infections (BSI) can be affected by a variety of factors including the collection technique to avoid contamination, the amount of blood volume collected, the timing of collection among other factors. Specifically, the early recognition of blood culture positivity and appropriate early source control are essential for successful treatment of patients with signs of a systemic response to the blood stream infection and end-organ dysfunction. Delay in recognition of blood culture positivity can lead to treatment delays along with possible disease progression.

Studies evaluated the usefulness of monocyte distribution width (MDW) for the assessment of emergency department patients with sepsis. It has been observed that monocyte activation in response to bacteremia leads to increased monocyte size. [5] MDW reflects a measure of a change in the size distribution of circulating monocytes. MDW has been evaluated for the aid of sepsis based on the definitions above. [6] The study by Crouser showed that the detection diagnosis of sepsis within 12 hours of ED presentation was aided when MDW was added. Similar, Polili et al found that the addition of MDW to the routine White Blood Cell (WBC) counts aids sepsis diagnosis and may be more useful than procalcitonin. [7]

It has not yet clearly established that MDW are elevated in bloodstream infections (BSI). BSI are diagnosed using blood cultures as gold standard for diagnosis. Blood cultures have a high sensitivity and specificity.[8] Up to thirty forty percent of septic shock patients will be blood culture positive and up to 25-30% negative for any type of culture. However, the diagnosis can take time delaying initiation of appropriate treatment. Additionally, in up to 50 % of cases BSI may be present without blood culture positivity due to the presence of uncultivable organisms or antibiotic treatment started prior to sampling.[9] MDW may be useful in not only aiding the diagnosis of sepsis but also in the expedited diagnosis of BSI.

This project will evaluate the usefulness of MDW for the diagnosis of blood culture positivity (BSI) in patients in the ED and reevaluate the usefulness of MDW in patients with BSI and sepsis. Consequently, if MDW indicate a high likelihood of bacteremia; antibiotic management in patients with suspected bacterial infections will be changed and aid appropriate antibiotic administration. On the other hand, a negative MDW test in the ED without additional risk factors or signs of infection (ie. Urinary tract, pneumonia, skin) or suspected severe sepsis or septic shock, patients may be treated supportively without use of antibiotics in the appropriate clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the Main Campus Emergency Department who had blood cultures ordered

Exclusion Criteria:

* Emergency Department Patients that do not have blood cultures ordered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Emergency Department patients older than 18 years with blood culture orders and blood culture blood draws.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Observed Sensitivity and Specificity of MDW >/= 20 U in Emergency Department Patients with Positive Blood Cultures | 09/2020 to 02/2023
Determine the negative predicative value of MDW assessments in Emergency Department patients at a cutoff threshold of <20 U in patients with negative blood cultures. | 09/2020 to 02/2023

OTHER OUTCOMES:
Exploratory Aim 1 Explore the sensitivity and specificity of MDW measurement in samples excluded due to the consideration of contaminated blood culture. Contaminants could be considered for BSI with skin flora or singular positive blood cultures. | 09/2020 to 02/2023
Exploratory Aim 2 Explore the sensitivity and specificity of MDW measurement in samples excluded due to use of antibiotics prior to the documented blood culture blood draw. | 09/2020 to 02/2023
Exploratory Aim 3a Explore changes in size of MDW from ED presentation to the last available measurement prior to discharge as sign of resolution of infection or sepsis/ measurement of treatment response. | 09/2020 to 02/2023
  When follow-up cultures are available the corresponding CBC MDW value should be below the cut-off of 20 U or at least 10 % reduced compared to when the blood cultures were positive. Chart review will be done to also evaluate the possibility of undiagnosed or nosocomial bacterial or viral co-infections such as urinary tract infections, pneumonia, abdominal infections as possible cause for continued elevated MDW. If MDW normalize in size and signs of infection are reduced this marker could be used to guide appropriate antibiotic therapy and early discontinuation of unnecessary antibiotic usage. This could lead to improved treatment strategies and reductions in emerging antibiotic resistance. If available, serial procalcitonin levels will be correlated with MDW values.
Exploratory Aim 3b Explore variations in MDW size on presentation based on reported symptom duration in Emergency Department patients. | 09/2020 to 02/2023
Exploratory Aim 4 Explore the value of MDW size at the time of hospital discharge is predictive for hospital readmission at day 28, day 30 or day 90 independent of infective cause. | 09/2020 to 02/2023
Exploratory Aim 5 Explore if MDW values are predictive SARS-CoV2 test or the need of admission for COVID-19 or influenza A/ B infection. | 09/2020 to 02/2023

CONTACTS AND LOCATIONS:
Overall Officials: Anja K Jaehne, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
We will not share individual subject data for privacy reasons. We plan to share aggregate data.

REFERENCES:
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; International Sepsis Definitions Conference. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Intensive Care Med. 2003 Apr;29(4):530-8. doi: 10.1007/s00134-003-1662-x. Epub 2003 Mar 28. PMID 12664219
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Lo RSL, Leung LY, Brabrand M, Yeung CY, Chan SY, Lam CCY, Hung KKC, Graham CA. qSOFA is a Poor Predictor of Short-Term Mortality in All Patients: A Systematic Review of 410,000 Patients. J Clin Med. 2019 Jan 8;8(1):61. doi: 10.3390/jcm8010061. PMID 30626160
- [Background] Crouser ED, Parrillo JE, Seymour C, Angus DC, Bicking K, Tejidor L, Magari R, Careaga D, Williams J, Closser DR, Samoszuk M, Herren L, Robart E, Chaves F. Improved Early Detection of Sepsis in the ED With a Novel Monocyte Distribution Width Biomarker. Chest. 2017 Sep;152(3):518-526. doi: 10.1016/j.chest.2017.05.039. Epub 2017 Jun 15. PMID 28625579
- [Background] Crouser ED, Parrillo JE, Martin GS, Huang DT, Hausfater P, Grigorov I, Careaga D, Osborn T, Hasan M, Tejidor L. Monocyte distribution width enhances early sepsis detection in the emergency department beyond SIRS and qSOFA. J Intensive Care. 2020 May 5;8:33. doi: 10.1186/s40560-020-00446-3. eCollection 2020. PMID 32391157
- [Background] Polilli E, Sozio F, Frattari A, Persichitti L, Sensi M, Posata R, Di Gregorio M, Sciacca A, Flacco ME, Manzoli L, Di Iorio G, Parruti G. Comparison of Monocyte Distribution Width (MDW) and Procalcitonin for early recognition of sepsis. PLoS One. 2020 Jan 10;15(1):e0227300. doi: 10.1371/journal.pone.0227300. eCollection 2020. PMID 31923207
- [Background] Opota O, Jaton K, Greub G. Microbial diagnosis of bloodstream infection: towards molecular diagnosis directly from blood. Clin Microbiol Infect. 2015 Apr;21(4):323-31. doi: 10.1016/j.cmi.2015.02.005. Epub 2015 Feb 14. PMID 25686695
- [Background] Fenollar F, Raoult D. Molecular diagnosis of bloodstream infections caused by non-cultivable bacteria. Int J Antimicrob Agents. 2007 Nov;30 Suppl 1:S7-15. doi: 10.1016/j.ijantimicag.2007.06.024. Epub 2007 Aug 17. PMID 17707613
- See also: Abstract — https://onlinelibrary-wiley-com.sladenlibrary.hfhs.org/doi/full/10.1111/acem.14906